CLINICAL TRIAL: NCT03441711
Title: The Utility of the sFlt-1/PlGF Ratio in Diagnosing Superimposed Preeclampsia and Predicting Adverse Outcomes in Subjects With Chronic Hypertension
Brief Title: sFlt-1:PlGF Ratio in Diagnosing Superimposed Preeclampsia
Status: Completed | Type: Observational
Sponsor: University of Tennessee (Other)
Responsible Party: Sponsor
Other Study IDs: 16-04377-XP
Record Dates: First submitted 2018-02-06; First posted 2018-02-22 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2019-01

CONDITIONS: Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — When blood sampling is clinically indicated, 10cc of maternal blood collected: at initial presentation, and at 2-7 d after initial, if undelivered.
  Lab analysis performed in batches: sFlt-1 level, PlGF level, & sFlt-1/PlGF ratio (for research purpose only at cost of investigators), post-collection of history, lab data, delivery data & outcomes.
  As clinically indicated (not altered for research purposes): Results for maternal urine-protein/creatinine ratio, CBC, CMP, LDH, & Uric acid will be collected.
  Ultrasound, performed by investigators for research purpose only, on weekly basis from the time of enrollment until delivery, to evaluate uterine artery Doppler, middle cerebral artery Doppler, umbilical artery Doppler, estimated fetal weight, & amniotic fluid volume.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1: elevated sFlt-1/PlGF ratio
- Group 2: normal sFlt-1/PlGF ratio

SUMMARY:
Preeclampsia: associated with poor placentation, incomplete uteroplacental spiral arteries remodeling. Result: ischemia, re-perfusion injury, oxidative stress.

A low-grade systemic inflammatory response is more pronounced in preeclampsia. This results in an imbalance between maternal circulating pro-angiogenic (PlGF & VEGF) & anti-angiogenic factors (sFlt-1).

PlGF & VEGF function as vasodilators & preserve structure & function of glomerular endothelium. sFlt-1 blocks these actions, resulting in hypertension, endothelial dysfunction & nephropathy.

Various stressors, including hypoxia, villous crowding, angiotensin II, & oxidative stress are associated with preeclampsia & mediate secretion of soluble vascular growth factor 1 (sVEGFR-1 or sFlt-1) by GADD45 (Growth Arrest and DNA Damage-45). GADD45 is one of a family of stress-induced genes sFlt-1 releases into maternal circulation. Excess sFlt-1 leads to endothelial dysfunction, hypertension & proteinuria.

Exogenously administered sFlt-1 results in syndrome of nephrotic range proteinuria, hypertension, and glomerular endotheliosis in animal models.

Women with preeclampsia tend to have higher sFlt-1 & lower PlGF, resulting in an increased ratio (sFlt-1:PlGF). The difference is greater in women who develop early-onset preeclampsia (before 34 wks gestation).

Verlohren, et al., showed an increased sFlt-1/PlGF ratio in patients with preeclampsia as compared to controls & patients with chronic/gestational hypertension.

Other work has examined the longitudinal changes in the individual values of sFlt-1 & PlGF over the course of the pregnancy, as well as the ratio.

Given the low prevalence of preeclampsia in the population, the positive predictive value remained low, however the negative predictive value approached 97% late in gestation. This suggests that the utility of the sFlt-1/PlGF may be in its ability to rule out preeclampsia.

More recently the PROGNOSIS study was designed to investigate the value of the sFlt-1/PlGF ratio for the prediction of the presence or absence of preeclampsia in the short term & found that a cutoff point of 38 for the sFlt-1/PlGF ratio is useful for predicting the short-term absence of preeclampsia in women with suspected disease (Negative predictive value 99.3% for ruling out preeclampsia within 1 week).

Hypothesis: In women with chronic hypertension, the sFlt-1/PlGF ratio will better predict the development of superimposed preeclampsia than clinical criteria alone.

DETAILED DESCRIPTION:
Subjects with a diagnosis of chronic hypertension made prenatally or in the first 20 weeks of pregnancy (+/- medical therapy). The clinical diagnosis of preeclampsia will follow the current criteria outlined by ACOG (American College of Obstetricians & Gynecologists) 10.

Study/Project Procedures:

* Blood draw at the time of initial presentation at the time of a clinically indicated blood draw (10cc maternal blood via venipuncture)
* Blood draw at 2-7 days after initial presentation if undelivered at the time of a clinically indicated blood draw(10 cc maternal blood via venipuncture)
* Laboratory analysis will be performed in batches after all clinical history, clinically indicated laboratory information, delivery information, and clinical outcomes recorded for sFlt-1 level, PlGF level, and the sFlt-1/PlGF ratio (not part of routine care and will be performed for research purposes only at the cost of the investigators).
* Urine protein creatinine ratio performed as clinically indicated (will not be altered for research purposes)
* Maternal CBC (Complete Blood Count), CMP (Complete Metabolic Profile), LDH (Lactate dehydrogenase), Uric acid as indicated clinically (will not be altered for research purposes)
* Ultrasound performed by the investigators for research purposes only evaluating the uterine artery Doppler, middle cerebral artery Doppler, umbilical artery Doppler, estimated fetal weight, and amniotic fluid volume on a weekly basis from the time of enrollment until delivery.
* Medical record abstraction of medical history, laboratory and clinical findings for both the mother and fetus.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age at enrollment: 20 0/7 weeks to 38 6/7 weeks gestation Pregnant women aged 14 to 45 years
* Presenting for admission for suspected superimposed preeclampsia
* Diagnosis of chronic hypertension made prenatally or in the first 20 weeks of pregnancy (+/- medical therapy)
* The clinical diagnosis of preeclampsia will follow the current criteria outlined by ACOG 10.

Exclusion Criteria:

* Age 45 years;
* Gestational age 19 6/7 weeks or less or 39 weeks or more ;
* Multiple gestations.

Ages: 14 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 150 pregnant subjects and their respective fetuses (total 300 subjects)
  Prospective cohort:
  * Group 1: elevated sFlt-1/PlGF ratio;
  * Group 2: normal sFlt-1/PlGF ratio.
Sampling Method: Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2016-02; Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
The diagnosis rate of superimposed preeclampsia for gestations of 20 0/7 weeks through 38 6/7 as evidenced by the degree of change in the 'sFlt-1/PlGF ratio' | From 20 0/7 weeks through 38 6/7 weeks.
  result at the point of enrollment; compared to the ratio result at 2-7 days post enrollment

SECONDARY OUTCOMES:
The diagnosis rate of Maternal morbidity HELLP syndrome for gestations of 20 0/7 weeks through 38 6/7 as evidenced by the degree of change in the 'sFlt-1/PlGF ratio' | between 20 0/7 weeks to 38 6/7 weeks gestation
  result at the point of enrollment; compared to the ratio result at 2-7 days post
The diagnosis rate of Eclampsia for gestations of 20 0/7 weeks through 38 6/7 as evidenced by the degree of change in the 'sFlt-1/PlGF ratio' | between 20 0/7 weeks to 38 6/7 weeks gestation
  result at the point of enrollment; compared to the ratio result at 2-7 days post
The diagnosis rate of Pulmonary edema for gestations of 20 0/7 weeks through 38 6/7 as evidenced by the degree of change in the 'sFlt-1/PlGF ratio' | between 20 0/7 weeks to 38 6/7 weeks gestation
  result at the point of enrollment; compared to the ratio result at 2-7 days post
The diagnosis rate of DIC (Disseminated Intravascular Coagulation) for gestations of 20 0/7 weeks through 38 6/7 as evidenced by the degree of change in the 'sFlt-1/PlGF ratio' | between 20 0/7 weeks to 38 6/7 weeks gestation
  result at the point of enrollment; compared to the ratio result at 2-7 days post
The diagnosis rate of Liver hematoma/rupture for gestations of 20 0/7 weeks through 38 6/7 as evidenced by the degree of change in the 'sFlt-1/PlGF ratio' | between 20 0/7 weeks to 38 6/7 weeks gestation
  result at the point of enrollment; compared to the ratio result at 2-7 days post
The diagnosis rate of Stroke for gestations of 20 0/7 weeks through 38 6/7 as evidenced by the degree of change in the 'sFlt-1/PlGF ratio' | between 20 0/7 weeks to 38 6/7 weeks gestation
  result at the point of enrollment; compared to the ratio result at 2-7 days post
The diagnosis rate of Death for gestations of 20 0/7 weeks through 38 6/7 as evidenced by the degree of change in the 'sFlt-1/PlGF ratio' | between 20 0/7 weeks to 38 6/7 weeks gestation
  result at the point of enrollment; compared to the ratio result at 2-7 days post

CONTACTS AND LOCATIONS:
Overall Officials: Giancarlo Mari, M.D., Principal Investigator — OB/GYN, MFM
Locations (1):
- Regional One Health Center for High Risk Pregnancies, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burton GJ, Jauniaux E. Placental oxidative stress: from miscarriage to preeclampsia. J Soc Gynecol Investig. 2004 Sep;11(6):342-52. doi: 10.1016/j.jsgi.2004.03.003. PMID 15350246
- [Background] Honigberg MC, Cantonwine DE, Thomas AM, Lim KH, Parry SI, McElrath TF. Analysis of changes in maternal circulating angiogenic factors throughout pregnancy for the prediction of preeclampsia. J Perinatol. 2016 Mar;36(3):172-7. doi: 10.1038/jp.2015.170. Epub 2015 Nov 19. PMID 26583938
- [Background] Xiong Y, Liebermann DA, Holtzman EJ, Jeronis S, Hoffman B, Geifman-Holtzman O. Preeclampsia-associated stresses activate Gadd45a signaling and sFlt-1 in placental explants. J Cell Physiol. 2013 Feb;228(2):362-70. doi: 10.1002/jcp.24139. PMID 22718299
- [Background] Redman CW, Sargent IL, Staff AC. IFPA Senior Award Lecture: making sense of pre-eclampsia - two placental causes of preeclampsia? Placenta. 2014 Feb;35 Suppl:S20-5. doi: 10.1016/j.placenta.2013.12.008. Epub 2014 Jan 11. PMID 24477207
- [Background] Maynard SE, Min JY, Merchan J, Lim KH, Li J, Mondal S, Libermann TA, Morgan JP, Sellke FW, Stillman IE, Epstein FH, Sukhatme VP, Karumanchi SA. Excess placental soluble fms-like tyrosine kinase 1 (sFlt1) may contribute to endothelial dysfunction, hypertension, and proteinuria in preeclampsia. J Clin Invest. 2003 Mar;111(5):649-58. doi: 10.1172/JCI17189. PMID 12618519
- [Background] Leanos-Miranda A, Campos-Galicia I, Isordia-Salas I, Rivera-Leanos R, Romero-Arauz JF, Ayala-Mendez JA, Ulloa-Aguirre A. Changes in circulating concentrations of soluble fms-like tyrosine kinase-1 and placental growth factor measured by automated electrochemiluminescence immunoassays methods are predictors of preeclampsia. J Hypertens. 2012 Nov;30(11):2173-81. doi: 10.1097/HJH.0b013e328357c0c9. PMID 22902831
- [Background] Verlohren S, Herraiz I, Lapaire O, Schlembach D, Moertl M, Zeisler H, Calda P, Holzgreve W, Galindo A, Engels T, Denk B, Stepan H. The sFlt-1/PlGF ratio in different types of hypertensive pregnancy disorders and its prognostic potential in preeclamptic patients. Am J Obstet Gynecol. 2012 Jan;206(1):58.e1-8. doi: 10.1016/j.ajog.2011.07.037. Epub 2011 Jul 30. PMID 22000672
- [Background] McElrath TF, Lim KH, Pare E, Rich-Edwards J, Pucci D, Troisi R, Parry S. Longitudinal evaluation of predictive value for preeclampsia of circulating angiogenic factors through pregnancy. Am J Obstet Gynecol. 2012 Nov;207(5):407.e1-7. doi: 10.1016/j.ajog.2012.08.010. Epub 2012 Aug 10. PMID 22981320
- [Background] Zeisler H, Llurba E, Chantraine F, Vatish M, Staff AC, Sennstrom M, Olovsson M, Brennecke SP, Stepan H, Allegranza D, Dilba P, Schoedl M, Hund M, Verlohren S. Predictive Value of the sFlt-1:PlGF Ratio in Women with Suspected Preeclampsia. N Engl J Med. 2016 Jan 7;374(1):13-22. doi: 10.1056/NEJMoa1414838. PMID 26735990